CLINICAL TRIAL: NCT01781494
Title: Immobilization Versus Immediate Motion After Anterior Submuscular Ulnar Nerve Transposition: Affect on Flexor-pronator Integrity
Brief Title: Immobilization Versus Immediate Motion After Anterior Submuscular Ulnar Nerve Transposition
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Kevin J. Renfree, Assistant Professor of Orthopedics, College of Medicine, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 11-001012
Record Dates: First submitted 2013-01-29; First posted 2013-02-01 (Estimated); Last update posted 2014-12-02 (Estimated); Status verified 2014-11

CONDITIONS: Cubital Tunnel Syndrome
MeSH Terms: conditions — Cubital Tunnel Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Immobilization (Active Comparator): Immobilization followed by protected range of motion
  Interventions: Procedure: Immobilization followed by protected range of motion
- Immediate range of motion (Experimental): Immediate motion after anterior submuscular ulnar nerve transposition
  Interventions: Procedure: Immediate range of motion

INTERVENTIONS:
Procedure: Immobilization followed by protected range of motion
  Arms: Immobilization
Procedure: Immediate range of motion
  Arms: Immediate range of motion

SUMMARY:
The goal of this study is to test the hypothesis that immediate elbow motion is safe after anterior submuscular ulnar nerve transposition, and will not result in disruption of the repaired flexor pronator origin, under which the nerve is placed. The advantages of immediate elbow motion after submuscular ulnar nerve transposition for performing activities of daily living and self-care are evident, however theoretical advantages include early "gliding" of the transposed ulnar nerve with a lower risk of nerve adhesions and subsequent traction neuritis, as well as improved blood flow and quicker, more complete, recovery of nerve function.

A group of 44 consecutive patients that are determined to be candidates for anterior submuscular ulnar nerve transposition based on history, positive findings on physical examination, and confirmatory electrodiagnostic testing will be prospectively randomized to either immediate motion or long arm cast immobilization after surgery. All patients will be counseled about the two postoperative treatment options (immobilization followed by protected range of motion versus immediate range of motion), risks involved with each treatment protocol, postoperative follow-up and need for radiographs. If they choose not to participate, they will be treated by the same postoperative protocol currently used by the principal investigator: arm sling at rest for six weeks with intermittent active assisted range of motion exercises.

ELIGIBILITY:
Inclusion Criteria:

* Candidates for anterior submuscular ulnar nerve transposition based on history, positive findings on physical examination, and confirmatory electrodiagnostic testing in Mayo Clinic Arizona

Exclusion criteria:

* Pregnancy
* Patients who have had prior ulnar nerve surgery
* Patients with other documented neurogenic processes identified on electrodiagnostic studies (ie: peripheral neuropathy, cervical radiculopathy, carpal tunnel syndrome)
* Workman's compensation patients
* Subluxing ulnar nerve
* Elbow contracture or stiffness
* Negative electrodiagnostic studies

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2014-01; Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
Change in the distance between the ligaclips on lateral elbow radiographs | Baseline to 3 months post-operatively

SECONDARY OUTCOMES:
Isokinetic strength testing of elbow flexion, forearm pronation, and wrist flexion | Baseline to 3 months post-operatively

CONTACTS AND LOCATIONS:
Overall Officials: Kevin Renfree, MD, Principal Investigator — Mayo Clinic